CLINICAL TRIAL: NCT07306195
Title: Comparison Between High and Low Level Para-aortic Lymphadenectomy in High and Intermediate Risk Endometrial Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmed Aouf (Other)
Responsible Party: Sponsor-Investigator, Ahmed Aouf, dr-sponsor, Kafrelsheikh University
Organization: Kafrelsheikh University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KFSIRB200-762
Record Dates: First submitted 2025-12-02; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Endometrial Cancer
Keywords: Endometrial Cancer; hystrectomy; para-aortic lymphadenectomy; high level para-aortic lymphadenectomy; low level para-aortic lymphadenectomy; survival outcome
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Intervention Model Description: This prospective, comparative clinical trial was conducted on 102 women diagnosed with high- or intermediate-risk EC , during the period from September 2022 to April 2025. The institutional review board (IRB) of Kafrelsheikh University approved the study. We complied with the ethical guidelines outlined in the Declaration of Helsinki throughout the study.The inclusion criteria consisted of women diagnosed with either intermediate- or high-risk EC, based on established pathological and radiological criteria.Eligible patients were stratified according to their risk category (intermediate or high risk) and subsequently randomized into two surgical groups based on the extent of PALD. Group A underwent high-level PALD, where lymphatic dissection was extended above the IMA up to the left renal vein. Group B underwent low-level PALD, in which lymph node dissection was confined to the inframesenteric region, extending from extending from the aortic bifurcation to just below the IMA.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The patient were randomized into two groups , group A and group B. The patients and the investigators were blinded from patient selection by giving the patient a sealed envelope . The patient allocation was done by computer software to achieve the randomization. The investigators were blinded from patient selection by handing them a sealed envelope and outcome assessors also were blinded from patient details at the follow up sessions
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A high (Active Comparator): underwent high-level PALD, where lymphatic dissection was extended above the IMA up to the left renal vein.
  Interventions: Procedure: high level para-aortic lymphadenectomy
- group B low (Active Comparator): underwent low-level PALD, in which lymph node dissection was confined to the infra-mesenteric region, extending from the aortic bifurcation to just below the IMA.
  Interventions: Procedure: low level para-aortic lymphadenectomy

INTERVENTIONS:
Procedure: high level para-aortic lymphadenectomy — All women underwent total hysterectomy with bilateral salpingo-oophorectomy combined with systematic pelvic lymphadenectomy and high-level PALD was done .The small bowel and mesentery were carefully mobilized to expose the aorta and inferior vena cava (IVC) above the IMA, with dissection proceeding cranially to the left renal vein. The anatomical landmarks were consistently identified to ensure complete lymphatic clearance within the defined field. Excised lymph nodes were counted intraoperatively and verified by histopathology.
  Arms: group A high
Procedure: low level para-aortic lymphadenectomy — All women underwent total hysterectomy with bilateral salpingo-oophorectomy combined with systematic pelvic lymphadenectomy and high-level PALD was done .The small bowel and mesentery were carefully mobilized to expose the aorta and inferior vena cava (IVC) , the dissection was restricted to the infra-mesenteric region between the aortic bifurcation and the IMA. The anatomical landmarks were consistently identified to ensure complete lymphatic clearance within the defined field. Excised lymph nodes were counted intraoperatively and verified by histopathology.
  Arms: group B low

SUMMARY:
Endometrial cancer (EC) is the most frequent gynecological malignancy in developed countries and ranks second in incidence worldwide after cervical cancer, accounting for nearly 10% of cancers in women . With the adoption of comprehensive surgical staging, the identification of extra-uterine disease has become central to treatment and prognosis. Lymph node involvement, particularly para-aortic nodal metastasis, represents one of the most important independent prognostic factors .

The uterus has a complex lymphatic drainage, with pathways leading to the obturator, iliac, caval, aortic, parametrial, and presacral basins. Direct channels from the uterine fundus to the para-aortic nodes via the infundibulopelvic ligament explain metastatic spread to the para-aortic region, although isolated para-aortic involvement in the absence of pelvic nodal disease is uncommon. Recognition of these drainage patterns underscores the importance of evaluating both pelvic and para-aortic lymph nodes in high- and intermediate-risk patients .

Several studies suggest that systematic lymphadenectomy, including the para-aortic region, improves survival by enhancing staging accuracy and guiding adjuvant therapy. Combined pelvic and para-aortic lymphadenectomy (PALD) has been associated with increased 5-year overall survival, improved disease-free survival, reduced recurrence, and decreased need for adjuvant radiotherapy . However, the optimal extent of para-aortic dissection remains debated. Para-aortic nodes are subdivided relative to the inferior mesenteric artery (IMA) into inframesenteric (low-level) and supramesenteric (high-level). While high-level PALD may improve detection of occult metastases, it increases surgical complexity and morbidity .

Risk stratification of EC guides the extent of staging. High-risk disease includes non-endometrioid histologies, grade 3 endometrioid carcinoma with >50% myometrial invasion, and advanced local spread. Intermediate-risk disease encompasses grade 1-2 tumors with deep or larger-volume myometrial invasion. Patients in these categories have a significant risk of nodal involvement (up to 16%), warranting para-aortic evaluation .

The present study aims to compare high versus low PALD in intermediate- and high-risk EC with emphasis on nodal yield, histopathological characteristics, staging, and oncological outcomes.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria consisted of women diagnosed with either intermediate- or high-risk EC, based on established pathological and radiological criteria. •Intermediate-risk patients included those with grade 1/2 endometrioid carcinoma with <50% myometrial invasion and tumor size >2 cm, grade 1/2 with 50-66% invasion, or grade 3 with <50% invasion.

  * High-risk cases were defined as non-endometrioid histology (serous or clear cell), grade 1 or 2 endometrioid carcinoma with more than 66% invasion, grade 3 with more than 50% invasion, or the presence of adnexal metastasis.

Exclusion Criteria:

* Patients were excluded if they had general contraindications to surgery, morbid obesity that precluded safe operative access, or if they declined to participate.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
descriptive operative outcome | 1 week
  The primary surgical outcome is para-aortic nodal yield
  how to measure paraaortic LN Yeild : surgical removal and pathological analysis, focusing on the number of nodes harvested (total yield) and the number of positive nodes (involved yield) relative to total nodes.

SECONDARY OUTCOMES:
survival outcome | 1 year
  Long-term oncological outcome, including (Overall survival) survival status at follow-up (alive, deceased, or lost to follow-up).

CONTACTS AND LOCATIONS:
Locations (1):
- Kafr Elsheikh University Hospital, Kafr ash Shaykh, Egypt

IPD SHARING:
Plan to Share IPD: Yes
there is a plan to make IPD available. It also means that a data dictionary (a description of the variables, or types of data, collected for each individual) will be provided so that the data can be fully interprete
Supporting Information: Study Protocol

REFERENCES:
- [Result] Somashekhar, S. P. et al. Prospective Non-randomized Control Trial on Role of Systematic High Para-Aortic Lymphadenectomy in Endometrial Cancer: Indian Study. Indian J Gynecol Oncolog 19, 6 (2021). 2. Jung, U. S., Choi, J. S., Bae, J., Lee, W. M. & Eom, J. M. Systemic Laparoscopic Para-Aortic Lymphadenectomy to the Left Renal Vein. JSLS 23, e2018.00110 (2019). 3. El-Agwany, A. S. & Meleis, M. H. Value and best way for detection of Sentinel lymph node in early stage endometrial cancer: Selective lymphadenectomy algorithm. European Journal of Obstetrics & Gynecology and Reproductive Biology 225, 35-39 (2018). 4. Petousis, S. et al. Combined pelvic and para-aortic is superior to only pelvic lymphadenectomy in intermediate and high-risk endometrial cancer: a systematic review and meta-analysis. Arch Gynecol Obstet 302, 249-263 (2020). 5. AlHilli, M. M. & Mariani, A. The role of para-aortic lymphadenectomy in endometrial cancer. Int J Clin Oncol 18, 193-199 (2013). 6. Zammarrelli, W. A. et al. Risk Stratification of Stage I Grade 3 Endometrioid Endometrial Carcinoma in the Era of Molecular Classification. JCO Precis Oncol e2200194 (2022) doi:10.1200/PO.22.00194. 7. Yang, Y., Wu, S. F. & Bao, W. Molecular subtypes of endometrial cancer: Implications for adjuvant treatment strategies. International Journal of Gynecology & Obstetrics 164, 436-459 (2024). 8. Thammineedi, S. R., Iyer, R. R., Naren, B. & Patnaik, S. C. Lymphadenectomy in Endometrial Cancers-A Review. Indian J Gynecol Oncolog 19, 77 (2021). 9. AlHilli, M. M. et al. Preoperative biopsy and intraoperative tumor diameter predict lymph node dissemination in endometrial cancer. Gynecologic Oncology 128, 294-299 (2013). 10. Hashmi, A. A. et al. Morphological Spectrum and Pathological Parameters of Type 2 Endometrial Carcinoma: A Comparison With Type 1 Endometrial Cancers. Cureus 12, (2020). 11. Song, S.-H. et al. Clinicopathologic Characteristics and Prognostic Factors of Stage I and II Endometrial cancer of the uter